CLINICAL TRIAL: NCT05748418
Title: Challenges Facing Community Health Workers (CHWs) in Provision of Health Services in Assiut Governorate
Brief Title: CHWs' Challenges and Job Satisfaction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doneez Amir Adly Eskander, Demonstrator, Assiut University
Other Study IDs: CHWs in Assiut Governorate
Record Dates: First submitted 2023-02-01; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Reproductive Issues

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
1. Determine the role of CHWs in health system.
2. Identify the barriers & obstacles they face in their work.
3. Determine factors related to motivation and satisfaction of CHWs job.
4. Identify the role of CHWs in family planning services.

DETAILED DESCRIPTION:
WHO consider "Community health workers should be members of the communities where they work, should be selected by the communities, should be answerable to the communities' needs and priorities, should be supported by the health system but not necessarily a part of the government and have shorter training than professional health workforce".

CHWs aims to provide appropriate, accessible care and bring care closer to mothers and babies, bridging the service delivery gap in underserved communities.

CHWs can effectively provide key primary, maternal, and newborn health care services including immunizations, tuberculosis treatment and contraceptive counseling.

CHWs face several challenges in reaching their full potential. Many of the obstacle's stem from a lack of understanding about their role within primary health system.

CHWs are faced by community and familial expectations of selflessness, equitably applied care, maintaining domestic responsibilities at home and implied understanding that extra work did not amount to extra pay.

In addition, motivation and satisfaction are key not only for retention but also for performance. Better workforce performance is positively associated with higher job satisfaction, and low levels of job satisfaction adversely affect employee commitment and sequentially affect achievement of organizational objectives and performance. Factors strongly associated with CHW satisfaction include relationships with health workers and communities, the availability of job aides and the capacity to provide services and with the training. On the other hand, CHWs were highly dissatisfied with the unavailability of transportation for carrying out their tasks and the lack of allowances or financial incentives. Also, Non-financial incentives include community recognition and respect, acquisition of valued skills, personal growth and development, accomplishment, peer support and community factors like relations with communities and leaders. Other supportive CHW programmed factors.

include frequent supervision and continuous training. therefore, CHW interventions must be implemented with an understanding of the complex challenges faced by CHWs and community members. This would in turn empower CHWs in navigating complex relationships within the community and the health system.

ELIGIBILITY:
Inclusion Criteria:

* Community health workers working in Assiut governorate.

Exclusion Criteria:

* Other healthcare providers.
* People with mental illness.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Community health workers working in Assiut governorate.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
CHWs' challenges | baseline
  challenges facing community health workers in provision of health services in Assiut governorate using self-administrated questionnaire.
CHWs' satisfaction | baseline
  Determine factors related to motivation and satisfaction of CHWs' job to achieve better performance using self-administrated questionnaire.

SECONDARY OUTCOMES:
role of community health workers in reproductive health services in Assiut governorate. | baseline
  Identify the role of CHWs in family planning services to to facilitate access to the service for its beneficiaries.

REFERENCES:
- [Background] Laurenzi CA, Skeen S, Rabie S, Coetzee BJ, Notholi V, Bishop J, Chademana E, Tomlinson M. Balancing roles and blurring boundaries: Community health workers' experiences of navigating the crossroads between personal and professional life in rural South Africa. Health Soc Care Community. 2021 Sep;29(5):1249-1259. doi: 10.1111/hsc.13153. Epub 2020 Sep 4. PMID 32885519
- [Background] Njororai F, Ganu D, Nyaranga KC, Wilberforce C. Role of Socio-Demographic and Environmental Determinants on Performance of Community Health Workers in Western Kenya. Int J Environ Res Public Health. 2021 Nov 8;18(21):11707. doi: 10.3390/ijerph182111707. PMID 34770222